CLINICAL TRIAL: NCT03606317
Title: Retrospective Review of Cachexia in Lung and Gastrointestinal Cancer Patients
Status: Active, not recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Parkland Health and Hospital System (Other)
Responsible Party: Principal Investigator, Anne Gilmore, Assistant Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU 092013-028
Record Dates: First submitted 2018-05-18; First posted 2018-07-30 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Cachexia
Keywords: Lung and gastrointestinal malignancies
MeSH Terms: conditions — Cachexia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The objective is to perform a retrospective chart review of patients with cachexia related to cancer in patients treated at UT Southwestern Medical Center and Parkland Hospital to evaluate the prognosis and practice patterns in management of cachexia and associated symptoms.

DETAILED DESCRIPTION:
The definition of cachexia has not been fully elucidated, but there are many similar parameters and guidelines associated with identifying patients with cachexia. Cachexia is a clinical diagnosis associated with weight loss, decreased muscle mass (sarcopenia), decreased strength, fatigue, and an increased inflammatory state. Patients with cachexia have a poorer prognosis than patients who have maintained their weight. Also, patients who have lost weight prior to initiating definitive therapy have worse side effects from subsequent therapy.

This study involves no treatment or invasive procedures. The chart review will attempt to characterize lung and gastrointestinal cancer related cachexia in the setting of a palliative care clinic including both primary treatment and treatment at the time of recurrence. Interventions in cachectic patients for weight control including nutritional support and supplements, pain control, anti-inflammatory medications, and appetite stimulants will be tracked along with clinical markers including weight and laboratory values.

ELIGIBILITY:
Inclusion Criteria:

Medical charts representing patients with a diagnosis of lung or gastrointestinal cancer with a tissue diagnosis from 1/1/2005 and onward treated at UT Southwestern or Parkland.

Exclusion Criteria:

There will be no absolute exclusion criteria as long as the inclusion criteria have been met.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects medical charts will be identified in the medical record data warehouses with diagnosis of lung or gastrointestinal cancer during the above time frame. Data from charts will be entered into a password protected excel spreadsheet. The charts will be identified by name, medical record number, and date of birth. These are all patients treated by all hospitals and clinics affiliated with the Parkland and UT Southwestern Health Systems. At the time of study, many of the patients will have expired but some will be alive and in the regional North Texas area. Thus, given the fact the majority of patients will have expired at the time of this study and the minimal risk nature of this retrospective chart review, we could not reasonably conduct this research with a full waiver of consent.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2013-11-26 (Actual); Primary Completion 2027-03-18 (Estimated); Study Completion 2027-03-18 (Estimated)

PRIMARY OUTCOMES:
Prognosis and practice patterns in the management of cachexia and its associated symptoms. | 10 years
  This study involves no treatment or invasive procedures. The chart review will attempt to characterize lung and gastrointestinal cancer related cachexia including both primary treatment and treatment at the time of recurrence. Interventions in cachectic patients for weight control including nutritional support and supplements, pain control, anti-inflammatory medications, and appetite stimulants will be tracked along with clinical markers, including weight and laboratory values.

CONTACTS AND LOCATIONS:
Overall Officials: Linda A Gilmore, Principal Investigator — University of Texas Southwestern Medical Center

IPD SHARING:
Plan to Share IPD: Undecided